CLINICAL TRIAL: NCT06014918
Title: A Smart Device Application for Acute Pain Service in Patients Undergoing Major Surgery: A Prospective Observational Feasibility Study
Brief Title: App for Acute Pain Service in Major Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hojin Lee, MD, Associate professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2304-053-1420
Record Dates: First submitted 2023-08-21; First posted 2023-08-28 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Mobile Applications; Pain, Postoperative; Smartphone; Patient Satisfaction
MeSH Terms: conditions — Pain, Postoperative; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: This study is designed to examine the feasibility of a smart device application to assess and manage postoperative pain in a single group of patients undergoing major surgery.
Masking Description: As this is an observational study to assess feasibility, the participants, care providers, researchers, and outcome assessors cannot be masked by the nature of the design.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients using a new application (Experimental): Patients will enter pain intensity and opioid analgesic side effects using a new application named 'Smart APS', developed for acute pain services, and later assess for adherence and satisfaction with the application use.
  Interventions: Device: A new smart device application (Smart APS)

INTERVENTIONS:
Device: A new smart device application (Smart APS) — The application sends alarms to patients to enter their pain intensity and opioid-related side effects at the times set by the researcher. Additional entries for severe pain or opioid side effects are also available at any other time. Researchers can monitor the results in real-time via an integrated web program. If a red flag sign is observed during regular office hours, an anesthesiologist participating in the research will visit the patient for assessment and intervention. In addition, patients can watch pre-made perioperative pain-related educational videos through the smart APS.

SUMMARY:
The app will be installed on the patient's smartphone before surgery. Patients will receive reminders to record their pain intensity and opioid-related side effects at the pre-determined time points until at least 2 days after surgery. The patient's compliance with the reminders will be assessed. On the second postoperative day, their satisfaction with pain control and app usage will be evaluated. Patients can also provide feedback on any issues they have encountered with the app during the study period.

DETAILED DESCRIPTION:
Following admission, the application will be installed on the enrolled patient's smartphone prior to surgery, and the patient will be instructed on the content of the program and how to use it. Educational videos within the app about postoperative pain control will be introduced to the patient at this time. At the pre-determined time points, until at least 2 days post-operatively, the patient will be reminded of the assessment via an alarm function and will enter post-operative pain intensity using an 11-point numeric rating scale or verbal rating scale and the presence of opioid-related side effects into the application. If a patient responds to the alarm 2 or more times per day, they will be considered to be compliant. Postoperative opioid consumption using patient-controlled analgesia and the amount of rescue analgesics will be assessed. Patients will be assessed with a survey on postoperative day 2 for overall satisfaction with pain control and usage of the application. Patients will also be able to provide feedback via the application or research staff on any errors or inconveniences they may have experienced while using the application throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 19 to 70 years who are scheduled for regular major surgery
* American Society of Anesthesiologists (ASA) physical status classification I or II
* Patients who are using a smartphone and are not expected to have any restrictions on application use

Exclusion Criteria:

* Unable to communicate
* Patients under the age of 19 and over the age of 70
* Patients who, in the opinion of the investigator or study staff, are not appropriate for this study

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-28 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-04-28 (Estimated)

PRIMARY OUTCOMES:
Patients' adherence rate to Smart APS | Postoperative day 1 and 2
  Proportion of patients who successfully used the smart APS among all patients.. Through Smart APS, a self-assessment is conducted three times a day, and it is assumed that the application has been used successfully if the patient completes an evaluation of pain intensity and opioid analgesic side effects at least twice on the first and second days after surgery.

SECONDARY OUTCOMES:
Patient satisfaction with pain management | Postoperative day 2
  Patient satisfaction with pain management using the 'Smart APS' app, rated on an 11-point scale (0 to 10 points, a higher number indicates higher satisfaction).
Patient satisfaction with application usage | Postoperative day 2
  A survey of patient satisfaction with the use of the 'Smart APS' app, consisted of 6 questions which are rated on a 7-point scale.

OTHER OUTCOMES:
Number of spontaneous assessments | Whole study period (from the day of surgery to at least 2 days after surgery)
  The number of spontaneous assessments made by the participant outside of the scheduled assessment time.
Amount of analgesics used | Whole study period (from the day of surgery to at least 2 days after surgery)
  Total volume of patient-controlled analgesia used and rescue analgesics.
Patient satisfaction with the provided audio-visual educational materials | Postoperative day 2
  Patient satisfaction with the provided four audio-visual materials is evaluated on a 0-10 scale. (A higher score indicates higher satisfaction)

CONTACTS AND LOCATIONS:
Overall Officials: Hojin Lee, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No